CLINICAL TRIAL: NCT05858541
Title: The Effects of Music Listening on Anxiety and Agitation in People With Mild and Moderate Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Assal Habibi, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APP-23-02029
Record Dates: First submitted 2023-04-28; First posted 2023-05-15 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Anxiety; Agitated Depression
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, and research staff involved in data collection and analysis will be masked to the assignment of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Listening (Experimental): Music Intervention - Music selection by LUCID The AI-based system for song selection responds to the collected measurement data (video and HRV) and music preference information (like/dislike button, music taste profile) to recommend the playlist for the listener. The songs are selected using 76 different musical features and raw audio information. The system uses these features to recommend and optimize recommendations for the listener. The video is only temporarily streamed from the device to extract a series of facial features to assist in music selection. This data stream is sent to the LUCID cloud platform via encrypted data in transit protocol; the facial features are extracted, and the video is deleted. The facial feature data, even when reconstructed, is not identifiable. No personally identifiable biometric measures are stored in LUCID servers at any time
  Interventions: Behavioral: Music Listening
- Audiobooks (Active Comparator): Audiobook selection A selection of 40 audiobooks spanning 4 genres (10 each from Literary Classics, Fantasy, Mystery, Non-fiction) will be available. For each session, the participant and their caregiver will be given a prompt to make a genre selection. After making the genre selection, one of the ten stories associated with that genre will be selected at random. All stories were sampled from the Audible audiobook database. Stories had to be 30 minutes in length to align with the length of the music interventions and the selected stories had to have had a 4- or 5-star rating to ensure quality.
  Interventions: Behavioral: Listening to Audiobooks

INTERVENTIONS:
Behavioral: Music Listening — The LUCID AI-based system for song selection responds to the collected measurement data (video and HRV) and music preference information (like/dislike button, music taste profile) to recommend the playlist for the listener. The songs are selected using 76 different musical features and raw audio information. The system uses these features to recommend and optimize recommendations for the listener
  Arms: Music Listening
Behavioral: Listening to Audiobooks — A selection of 40 audiobooks spanning 4 genres (10 each from Literary Classics, Fantasy, Mystery, Non-fiction) will be available. For each session, the participant and their caregiver will be given a prompt to make a genre selection. After making the genre selection, one of the ten stories associated with that genre will be selected at random. All stories were sampled from the Audible audiobook database. Stories had to be 30 minutes in length to align with the length of the music interventions and the selected stories had to have had a 4- or 5-star rating to ensure quality.
  Arms: Audiobooks

SUMMARY:
Advancing age is associated with an increased risk of developing dementia which can lead to a rapid acceleration in both the healthcare costs and caregiver burden. There is a need to develop non-pharmacological and easily accessible modalities of support for the well-being and enhancing quality of life for individuals with dementia. There is evidence that music listening is associated with stress and anxiety reduction in older adults. Here, the investigators aim to assess the effects of music listening as provided by a novel digital music-based intervention (developed by LUCID) on mood, anxiety, and quality of life in individuals at the early stages of dementia. LUCID uses reinforcement learning machine learning to curate and personalize the musical playlist while incorporating monoaural theta auditory beat stimulation (ABS) into the music. The study will be conducted remotely with study hardware (tablets and Bluetooth speakers) being delivered to caregivers/participants. The study will take place over an 8- week period, with participants completing four 30 mins music or audiobook listening sessions per week. Pre and post-intervention assessments will be done via Zoom with the presence of a research staff member. The control condition consists of a randomized list of short audiobooks. The experimental condition consists of music and monoaural ABS curated by LUCID's AI system. The investigators hypothesize that the LUCID AI music curation system, compared to audiobooks, will be correlated with a greater reduction in measures of anxiety and agitation and an enhancement of mood and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Mild to Moderate Cognitive Impairment (mild: MOCA scores (18-25); moderate: MOCA scores (10-17))
* Aged 65-85.

Exclusion Criteria:

* Unmanaged hearing loss (defined as the average pure-tone average threshold of 35 dB HL or greater without the use of hearing instruments or personal sound amplification product) - self-report
* Severe Tinnitus
* Hyperacusis
* Current (but not prior) severe psychiatric disorder, an unstable or serious medical condition that may limit participation in the assessments.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Agitation Trait | 8 weeks
  Change in agitation as measured by the Cohen-Mansfield Agitation Index
Agitation State | pre and post 20 mins session for a total of 32 sessions
  Change in agitation as measured by Overt Agitation Scale (OAS)
Agitation State | pre and post 20 mins session for a total of 32 sessions
  Change in agitation as measured by Positive and Negative Syndrome Scale, Excited Component (PANSS-EC)

SECONDARY OUTCOMES:
Anxiety | 8 weeks
  Change in Anxiety in Dementia Scale (RAID)-Minimum value: 0, Maximum value: 54. Higher score
Anxiety | 8 weeks
  Change in State-trait cognitive and somatic anxiety (STICSA)

OTHER OUTCOMES:
Depression | 8 weeks
  Change in depression as measured by Geriatric Depression Scale 0 is minimum and 15 is maximum with 15 being highest rate of depression
Well-being | 8 weeks
  Change in quality of life as measured by Cornell Brown Scale for Quality of Life in Dementia - Minimum score: -38. Maximum score: 38. Higher score indicates better outcome (increased quality of life)
Caregiver Burden | 8 weeks
  Change in caregiver burden measured by Zarit caregiver burden
Anxiety and Mood | pre and post 20 mins session for a total of 32 sessions
  Change in Mood and Anxiety as measured by PANAS Positive and Negative Affect Schedule
Arousal | pre and post 20 mins session for a total of 32 sessions
  Change in affect as measured by high low arousal
Valence | pre and post 20 mins session for a total of 32 sessions
  Change in affect as measured by positive negative valence
Memory | 8 weeks
  Changes in memory recall measured by vividness and specificity of recalled memories

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data and protocol will be available upon completion of the data and analysis